CLINICAL TRIAL: NCT01980290
Title: Observational Multicenter Study in Ex-People Who INject Drugs (Ex-PWIDs) to Evaluate Efficacy, Safety, and Adherence to TElaprevir in Combination With Pegylated Interferon Alfa and Ribavirin in Genotype 1 ChRonic HepATitis C PatiEnts
Brief Title: Telaprevir With Peginterferon Alfa & Ribavirin in Ex-People Who INject Drugs Infected by Genotype 1 Chronic Hepatitis C
Acronym: INTEGRATE
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100966; VX-950HPC4017 (Other: Janssen Pharmaceutica NV - CTMS ID)
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis, Chronic
Keywords: HCV genotype 1; Liver Fibrosis; ex-People who INject Drugs (ex-PWIDs)
MeSH Terms: conditions — Hepatitis, Chronic; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect information on the efficacy, safety and tolerability of telaprevir (in combination with other medications), in patients who have a history of intravenous drug use with genotype 1 chronic hepatitis C, under substitution therapy (eg., methadone, buprenorphine) and/or followed in addiction centres.

DETAILED DESCRIPTION:
This is a multicenter, non-interventional, observational, prospective study to evaluate the efficacy, safety, and adherence to telaprevir in ex-People Who Inject Drugs (ex-PWIDs) infected with genotype 1 chronic hepatitis C and any fibrosis stage including compensated cirrhosis, who are receiving substitution therapy (eg, methadone, buprenorphine) and/or are being followed in an addiction center. Patients may be treatment naïve or relapsers. Participating physicians are to offer enrollment in this study to all eligible patients at their site in who they plan to initiate triple therapy with telaprevir, pegylated interferon alfa (PegIFN alfa), and ribavirin (RBV). A target of 115 patients will participate in this study. The duration of each patient's participation in this study will be up to approximately 60 weeks. After obtaining the signed participation agreement or ICF, selection criteria will be reviewed to verify the patient's eligibility. Data will be recorded in the electronic case report form (CRF) at 6 time points for each patient which correspond to routine care visits: inclusion, and at the patient's routine care visit closest to Week 4, 12, and 24, end of treatment, and end-of-follow-up (e.g., approximately 12 weeks after end-of-treatment). No additional blood, urine, or other biological samples will be required, and no additional investigations, beyond the routine clinical management of the patient, will be performed.

ELIGIBILITY:
Inclusion Criteria:

Have HCV genotype 1, a quantifiable serum HCV RNA, recent (within 18 months of baseline) documentation of the degree of liver fibrosis (Metavir F0-F4; Ishak 0-6) assessed by liver biopsy or non-invasive test (eg, fibrotest, fibroscan); Physician decision to start triple therapy with telaprevir and PegIFN alfa/RBV; Have never been treated with antiviral treatment (naïve) or who have relapsed after IFN or PegIFN plus RBV (relapsers); History of injecting drugs and are currently under stable substitution therapy (eg, methadone, buprenorphine) and/or followed in an addiction center.

Exclusion Criteria:

Infected or coinfected with HCV of a genotype other than genotype 1; Previous or current treatment with a DAA therapy; Have any contraindication specified in the SmPC for telaprevir, PegIFN alfa, or RBV; Have a history or other evidence of decompensated liver disease, or have coinfection with active hepatitis B or HIV; Currently participating in another investigational study or clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men or women who have HCV infection genotype 1, a quantifiable serum HCV RNA, documentation of the degree of liver fibrosis assessed by liver biopsy or non-invasive test (eg, fibrotest, fibroscan), physician decision to start triple therapy with telaprevir and PegIFN alfa/RBV, have never been treated with antiviral treatment (naïve) or who have relapsed after IFN or PegIFN plus RBV (relapsers), have a history of injecting drugs, and are currently under stable substitution therapy (eg, methadone, buprenorphine) and/or followed in an addiction center will be eligible to enter this study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Sustained Virologic Response at 12 weeks (SVR12) | Week 12
  HCV RNA <25 IU/mL, at 12 weeks (SVR12) after the last dose of anti-HCV treatment (telaprevir, PegIFN alfa, RBV)

SECONDARY OUTCOMES:
adherence to telaprevir until Week 12 | week 12
  adherence as measured by pill count and/or patient questionnaire (modified medication adherence self-report inventory [M-MASRI]
adherence to PegIFN alfa and RBV | at end of treatment (week 24)
  adherence as measured by pill/vial count and/or patient questionnaire (M-MASRI)
on-treatment virologic response undetectable | week 12 and end of treatment ()
  rapid virologic response [RVR] and extended rapid virologic response [eRVR], Week 12, end of treatment) based on viral load, as measured by HCV RNA <25 IU/mL undetectable
on treatment virologic response | week 12 and end of treatment ()
  rapid virologic response [RVR] and extended rapid virologic response [eRVR], Week 12, end of treatment) based on viral load, as measured by HCV RNA <25 IU/mL
health-related quality of life based on EQ-5D | on day 1 and routine visits closest to week 4, 12, 24 and end of treatment and end of follow-up (up to approximately 60 weeks)
  The EQ-5D consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take 1 of 3 responses. The responses record 3 levels of severity (no problems/some or moderate problems/extreme problems). A standard vertical 20 cm visual analogue scale (similar to a thermometer) for recording an individual's rating for their current health-related quality of life state is also included ranging from 0 (worst imaginable health state) to 100 (best imaginable health state)
Hospital Anxiety and Depression Scale (HADS) | on day 1 and routine visits closest to week 4, 12, 24 and end of treatment and end of follow-up (up to approximately 60 weeks)
  HADS is a validated 14-item scale with 7 of the items relating to anxiety and 7 relating to depression. Each item is scored from 0 to 3, with higher scores indicating greater likelihood of depression or anxiety. Cases of anxiety or depression are each defined by subscale scores of 8 or greater, and categorized as normal (score of 0-7), mild (score of 8-10), moderate (score of 11-14), and severe (score of 15-21). The recall period is the past week.
alcohol use disorders identification test (AUDIT) | on day 1 and routine visits closest to week 4, 12, 24 and end of treatment and end of follow-up (up to approximately 60 weeks)
  The AUDIT questionnaire consists of 10 questions about a patient's quantity and frequency of alcohol use. The response to 8 of the questions are scored as 0 = never, 1 = monthly or less, 2 = 2 to 4 times a month, 3 = 2 to 3 times a week, 4 = 4 or more times a week. Two questions are scored as 0 = no, 2 = yes, but not in the last year, 4 = yes, during the last year. A score of 8 or more is associated with harmful or hazardous drinking

CONTACTS AND LOCATIONS:
Locations (18):
- Belgium (4):
  - Antwerp
  - Brussels
  - Genk
  - Haine-Saint-Paul
- France (3):
  - Lomme
  - Montpellier
  - Perpignan
- Germany (5):
  - Berlin
  - Biberach
  - Kassel
  - München
  - Münster
- Maastricht, Netherlands
- Switzerland (2):
  - Lausanne
  - Zurich
- United Kingdom (3):
  - Dundee
  - London
  - Nottingham

REFERENCES:
- [Derived] Robaeys G, Christensen S, Lucidarme D, Arain A, Bruggmann P, Kunkel J, Keim S, Jakel M, DeMasi R, Liu C, Lonjon-Domanec I, Foster GR. Chronic Hepatitis C Treatment in Patients with Drug Injection History: Findings of the INTEGRATE Prospective, Observational Study. Infect Dis Ther. 2017 Jun;6(2):265-275. doi: 10.1007/s40121-017-0158-x. Epub 2017 May 5. PMID 28477061